CLINICAL TRIAL: NCT07300163
Title: Foot Temperature and Diabetic Foot Ulcer Risk: Using the FeetSee Device to Generate a Unique Foot Temperature Dataset.
Brief Title: FeetSee Thermal Images Collection Protocol in Diabetes Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Diabetis JSC (Industry)
Collaborators: Horizon 2020 - European Commission (Other); Manchester University NHS Foundation Trust (Other Government); Lancashire Teaching Hospitals NHS Foundation Trust (Other); Vilnius University Hospital Santaros Klinikos (Other)
Responsible Party: Sponsor
Other Study IDs: FS-HRA_01-PR; RAS ID [345382] (Other: The Integrated Research Application System (IRAS) , UK); 10-036-T-0004 (Other Grant/Funding Number: European Horizon Programme)
Record Dates: First submitted 2025-12-10; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- FeetSee Foot Monitoring Cohort: Adults with type 1 or type 2 diabetes, peripheral neuropathy, and a recently healed plantar diabetic foot ulcer will use the FeetSee System at home in addition to their usual diabetic foot care. After baseline clinical assessment and training, participants will be asked to acquire at least one thermal (and accompanying optical) image of the plantar surface of both feet per day using the FeetSee thermal camera, stand, and smartphone/tablet application over the follow-up period (approximately 6-9 months) or until a new diabetic foot ulcer develops. Images are uploaded securely for later analysis of plantar temperature patterns. No experimental drug or change in standard clinical management is mandated by the protocol; the device is used for image collection only.
  Interventions: Device: FeetSee thermal camera

INTERVENTIONS:
Device: FeetSee thermal camera — The FeetSee Device consists of: (1) a smartphone/tablet-connected thermal imaging camera, (2) a mobile application installed on the participant's own mobile device, and (3) a stand to hold the device in a fixed position for imaging. Participants are instructed to take at least one bilateral plantar thermal and optical image of their feet per day at home over 6-9 months. Images are securely uploaded to cloud storage. The device is used for thermal image collection and is not a replacement for standard diabetic foot self-examination and routine clinical foot care; no treatment decisions are mandated by the study protocol.

SUMMARY:
Diabetic foot ulcers (DFUs) are a major cause of morbidity, lower-extremity amputation and healthcare costs in people with diabetes. DFUs often develop without pain or warning symptoms because of diabetic peripheral neuropathy, so patients may not recognise early signs of tissue damage. Monitoring plantar foot skin temperature is a promising strategy to detect early "hot-spots" of inflammation that precede ulceration and could trigger timely preventive action.

This prospective, single-group study will enrol adults with type 1 or type 2 diabetes, a history of plantar DFU that has been healed for at least 6 weeks, and evidence of diabetic peripheral neuropathy. Participants will be recruited from hospital clinics in the United Kingdom and Lithuania. After a baseline assessment (including medical history and neuropathy testing), each participant will receive the FeetSee system, consisting of a thermal camera attached to their own smartphone or tablet, a stand, and the FeetSee mobile application.

Participants will be instructed to acquire thermal and optical images of both feet at home at least once per day for 6-9 months, or until a new DFU develops. Images will be uploaded securely to cloud storage, where the FeetSee algorithm will analyse temperature patterns, comparing mirrored regions of both feet to identify potential inflammatory "hot-spots" associated with DFU risk. Participants will continue to receive standard clinical care throughout the study.

The primary objective is to generate a longitudinal foot temperature dataset in this high-risk population and use it to retrospectively test and refine the FeetSee algorithm for predicting DFU occurrence. The primary outcome is the incidence of new DFUs during follow-up. Secondary objectives are to assess the feasibility and acceptability of daily device use (recruitment, retention, adherence, user and healthcare-provider questionnaires) and to document any device-related or system-related safety issues.

DETAILED DESCRIPTION:
This is a prospective observational study with a single cohort of approximately 100 adults with type 1 or type 2 diabetes and a recently healed plantar DFU, conducted at hospital sites in the United Kingdom and at Vilnius University Hospital Santaros Klinikos in Lithuania. Eligibility requires peripheral neuropathy (defined by abnormal 10 g monofilament and/or vibration perception threshold testing) and at least one palpable foot pulse. Key exclusions include active DFU, active Charcot neuro-osteoarthropathy, severe peripheral arterial disease (no palpable foot pulses), major lower-limb amputation above the metatarsophalangeal joints, and medical or cognitive conditions that would prevent safe use of the device.

After informed consent and baseline assessments, participants are trained to use the FeetSee thermal camera, stand, and smartphone/tablet app at home. They are asked to remove footwear and socks and keep their feet non-weight-bearing for about 10 minutes before each measurement, then acquire at least one bilateral plantar image per day. Study staff provide intensive technical support during the first week and then schedule telephone check-ins approximately every three weeks, with additional troubleshooting as needed. Adherence is monitored via device-logged usage; failure to use the device for 21 consecutive days is considered loss to follow-up.

Thermal images are pseudo-anonymised and transferred securely to cloud infrastructure, where the FeetSee algorithm uses an active-shape model to detect foot contours and compares mirrored plantar regions for temperature differences above a predefined threshold (e.g.,>2.2 °C), indicative of local inflammation. The analyses performed by the device manufacturer (Diabetis JSC) will use the resulting temperature maps and clinical outcomes to estimate the sensitivity and specificity of the current algorithm for predicting incident DFUs and to develop refined algorithms. All other clinical and questionnaire data are analysed by the academic research team.

Feasibility outcomes include recruitment rate, retention, frequency of device use, and the number and nature of technical support contacts. Acceptance of the technology by both patients and healthcare professionals is assessed with questionnaires based on the Unified Theory of Acceptance and Use of Technology (UTAUT), covering performance expectancy, effort expectancy, social influence, facilitating conditions, self-efficacy, attitudes toward FeetSee, technology anxiety, and perceptions of personal DFU risk. Safety outcomes include the collection and classification of any adverse events and the identification of any device-related problems.

ELIGIBILITY:
Inclusion Criteria:

* Males/females aged over 18 years.
* Type 1 or type 2 diabetes.
* History of plantar diabetic foot ulcer(s).
* Foot ulcer healed for at least 6 weeks before entry into study, as determined by a specialist healthcare provider.
* Presence of diabetic peripheral neuropathy defined by either of the following:

  * Inability to detect the monofilament (10g) applied at two foot sites, including the apex of the Hallux (ADA guidelines 2008 Diabetes Care 31(1)).
  * A Vibration Perception Threshold (VPT) >20V, and/or by inability to detect application of the monofilament at the apex of the Hallux.
* Presence of at least one palpable foot pulse.

Exclusion Criteria:

* Active foot ulceration.
* Active Charcot neuro-osteoarthropathy.
* Severe vascular disease (complete absence of any foot pulses).
* Lower limb/foot amputation greater than metatarsophalangeal disarticulation.
* Active malignancy, immunosuppressive disease.
* Physical or mental condition(s) that limit the ability to follow instructions for the study, based on clinical judgment by the physician, such as inability to use the device without assistance.
* Current participation in another clinical investigation of a medical device that is contraindicated for either study procedure/outcome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (≥18 years) with type 1 or type 2 diabetes, a history of plantar diabetic foot ulcer(s) that have been fully healed for at least 6 weeks, clinical evidence of diabetic peripheral neuropathy, and at least one palpable foot pulse. This is a high-risk population for recurrent plantar diabetic foot ulceration, without active ulceration, active Charcot neuro-osteoarthropathy, severe peripheral arterial disease, or major lower-limb amputation (above metatarsophalangeal disarticulation).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-12-10 (Estimated); Primary Completion 2027-05-30 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
DFU occurrence over the six to nine-month follow-up period. | From baseline (enrolment) until study completion or development of a new DFU, up to 9 months per participant.
  Proportion of enrolled participants who develop at least one new plantar diabetic foot ulcer (DFU) during the study follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Neil Reeves, Prof, Phd, Principal Investigator — Manchester University NHS Foundation Trust (MFT); Loretta Vileikyte, Prof, MD, Principal Investigator — Lancashire Teaching Hospitals NHS Foundation Trust
Locations (3):
- Vilnius University Hospital Santaros Klinikos, Vilnius, Lithuania
- United Kingdom (2):
  - Lancashire Teaching Hospitals NHS Foundation Trust, Lancaster
  - Manchester University NHS Foundation Trust (MFT), Manchester